CLINICAL TRIAL: NCT05783258
Title: Comparative Evaluation of the Coronally Advanced Flap (CAF) Using a Connective Tissue Graft From the Tuberosity (tCTG) or L-PRF Membranes: a Randomized Controlled Clinical Trial.
Brief Title: Connective Tissue Graft From Tuberosity Area and L-PRF Associated With Coronally Advanced Flap for Root Coverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Michele Paolantonio, Full time professor, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13032023
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Gingival Recession
Keywords: Root coverage; Periodontal plastic surgery
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAF+tSCTG (Experimental): 15 sites will be treated.The extent of the depth of the recession will be reported on the anatomical papillae and, after adding 1 mm, 2 horizontal incisions of approximately 3 mm will be made at the base of the surgical papillae laterally to the recession.Two divergent releasing incisions will be made extending approximately 2-3 mm into the alveolar mucosa.The surgical papillae will be detached in partial thickness. A full thickness dissection will be performed from the bottom of the recession to expose approximately 3mm of the crest bone.A partial thickness dissection will be performed in the most apical portion of the flap until complete passivation of the flap is obtained.The harvesting of the epithelial-connective graft will be performed at the level of the maxillary tuberosity. The de-epithelialised graft will be sutured at the level of the de-epithelialised anatomical papillae.The flap will be repositioned coronally suturing the anatomical papillae on the surgical ones.
  Interventions: Procedure: Periodontal surgery with CAF+tSCTG
- CAF+L-PRF (Active Comparator): 15 sites will be treated.The extent of the depth of the recession will be reported on the anatomical papillae and, after adding 1 mm,2 horizontal incisions of approximately 3 mm will be made at the base of the surgical papillae laterally to the recession. Two divergent releasing incisions will be made extending approximately 2-3 mm into the alveolar mucosa. The surgical papillae will be detached in partial thickness. A full thickness dissection will be performed from the bottom of the recession to expose approximately 3mm of bone.A partial thickness dissection will be performed in the apical portion of the flap to obtain complete passivation.The L-PRF membranes will be realized centrifuged venous blood collected in two 10-ml sterile tubes at 3000 rpm for 10 minutes and squeezing the fibrin clot. L-PRF membranes will be superimposed to crete a double layer of about 2 mm thickness.The flap will be repositioned coronally suturing the anatomical papillae on the surgical ones.
  Interventions: Procedure: Periodontal surgery with CAF+L-PRF

INTERVENTIONS:
Procedure: Periodontal surgery with CAF+tSCTG — Coronally advanced flap and subepithelial connective tissue graft harvested from the maxillary tuberosity area.
  Arms: CAF+tSCTG
Procedure: Periodontal surgery with CAF+L-PRF — Coronally advanced flap and L-PRF membranes
  Arms: CAF+L-PRF

SUMMARY:
The aim of the present randomized controlled clinical study is to compare the efficacy of subepithelial connective tissue graft harvested from the maxillary retromolar tubeosity area and L-PRF membranes in the treatment of RT1 recessions by coronally advanced flap.

A total of 30 patients will be recruited and randomly assigned to the test group treated with CAF+tSCTG or the control group treated with (CAF+L-PRF). For each experimental site the parameters of gingival recession (GR), pocket depth (PD), clinical attachment level (CAL), keratinized gingiva width (KT) and gingival thickness (GT) will be analyzed at baseline (T0) and at 12 months after the surgical procedure (T1). In addition, was also evaluated the different morbidity of the two surgical techniques, using the VAS scale values recorded in the first 2 weeks following surgery. It was checked the Patient Related Esthetic Score and Dentine hypersensivite reduction.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a class RT1 recession;
* age > 18 years;
* systemic health conditions that do not affect the periodontium;
* Non smoker;
* FMPS and FMBS values < 20% before the surgical procedure;
* absence of implants or subgingival restorations in the sites to be treated;
* presence of adequate tissue distal to the last maxillary molar.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-10-29 (Actual); Study Completion 2023-10-29 (Actual)

PRIMARY OUTCOMES:
Gingival thickness | 12 months
  Gingival tissue thickness 2 mm apical to the recession

SECONDARY OUTCOMES:
Keratinized tissue height | 12 months
  Distance between gingival margin and Mucogingival Junction
Gingival recession | 12 months
  Distance from cementoenamel junction and gingival margin
Complete root coverage | 12 months
  Percentage of experimental sites that achieved complete root surface coverage.
Clinical attachment level | 12 months
  Distance between cementoenamel junction(CEJ) and depth of the pocket
Pocket depth | 12 months
  Distance between gingival margin and bottom of the pocket

CONTACTS AND LOCATIONS:
Locations (1):
- Michele Paolantonio, Pescara, Italy

IPD SHARING:
Plan to Share IPD: No